CLINICAL TRIAL: NCT00330863
Title: Preventing Relapse: Oral Antipsychotics Compared To Injectables: Evaluating Efficacy (PROACTIVE)
Brief Title: Preventing Relapse in Schizophrenia: Oral Antipsychotics Compared To Injectables: Evaluating Efficacy
Acronym: PROACTIVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01MH070007-01 (NIH); U01MH070007-01 (NIH); U01MH070023 (NIH); U01MH070011 (NIH); U01MH070009 (NIH); U01MH070008 (NIH); U01MH070017 (NIH); U01MH070010 (NIH); U01MH070016 (NIH); U01MH070012 (NIH); DSIR 83-ATAP (Other Grant/Funding Number: National Institute of Mental Health)
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Relapse; Prevention; Schizophrenia; Injectable Medication
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Recurrence | interventions — Risperidone; Olanzapine; Quetiapine Fumarate; ziprasidone; Aripiprazole; Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Injectable (Experimental): Participants assigned to receive long-acting injectable risperidone
  Interventions: Drug: Risperidone microspheres
- Oral (Active Comparator): Participants assigned to receive oral "atypical" antipsychotic medication
  Interventions: Drug: Risperidone; Drug: Olanzapine; Drug: Quetiapine; Drug: Ziprasidone; Drug: Aripiprazole; Drug: Paliperidone

INTERVENTIONS:
Drug: Risperidone microspheres — Minimum dose is 12.5 mg every 2 weeks. Maximum dose is 75 mg every 2 weeks.
  Other Names: Risperdal Consta
  Arms: Injectable
Drug: Risperidone — Target dose is 4 mg/day.
  Other Names: Risperdal
  Arms: Oral
Drug: Olanzapine — Target dose is 15 mg/day.
  Other Names: Zyprexa
  Arms: Oral
Drug: Quetiapine — Target dose is 600 mg/day.
  Other Names: Seroquel
  Arms: Oral
Drug: Ziprasidone — Target dose is 120 mg/day.
  Other Names: Geodon
  Arms: Oral
Drug: Aripiprazole — Target dose is 20 mg/day.
  Other Names: Abilify
  Arms: Oral
Drug: Paliperidone — Target dose is 6 mg/day.
  Other Names: Invega
  Arms: Oral

SUMMARY:
This study is designed to find out whether taking antipsychotic medication once every two weeks by injection compared to taking daily oral medication will help people with schizophrenia maintain better control of their symptoms.

DETAILED DESCRIPTION:
As is the case with many chronic illnesses, it can be challenging for people with schizophrenia to take multiple pills every day on a long-term basis. At the same time, missing or discontinuing the anti-psychotic medications that treat schizophrenia substantially increases the risk of relapse and re-hospitalization. This study will determine how effective long-acting injectable risperidone is compared to oral antipsychotic medications to help patients who have schizophrenia. Patients who enroll in the study will be randomly assigned to receive either long-acting injectable risperidone or to receive oral "atypical" antipsychotic medication. The "atypical" antipsychotics that are included for patients in the oral group are: aripiprazole, olanzapine, quetiapine, risperidone, and ziprasidone. Patients in the "oral" group will receive whichever of the five "atypical" antipsychotic medications they and their study doctor decide is best for them. Patients in the "oral" group will be allowed to switch to others of the five medications during the study if they and their doctor think that is best.

Patients in this study will be evaluated at the beginning of the study and then again every two weeks for up to 30 months (2 1/2 years). Each two-week visit will take about 20 minutes. At the visit, patients will receive medication and will be examined for side effects of the medications, their vital signs (heart rate, blood pressure, weight, and waist measurement) will be measured, and they will be asked a few questions about attendance at visits and taking medication. The visit that occurs every three months will take about one hour, instead of 20 minutes, and will include additional questions, an examination for muscle stiffness or abnormal body movements, and an interview from a member of the research team conducted using computer technology. In addition, blood and urine samples may be collected about seven times throughout the 30 months of the study treatment. Patients who enroll in this study after the halfway point of the study, may not receive a full 30 months of treatment, but it is planned that all patients will have the opportunity to receive no less than 18 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* All schizophrenia and schizoaffective patients whose clinicians are considering long-term treatment with an "atypical" (second generation) antipsychotic medication
* Worsening of illness (schizophrenia) within 12 months of study entry as defined by: hospitalization, increased level of clinical care, and/or present clinical Global Impressions Severity rating of moderate or worse

Exclusion Criteria:

* First episode patients as defined by a patient who: has never received antipsychotic medication and has never been hospitalized for psychiatric illness; or, is receiving antipsychotic medication for the first time associated with a first diagnosis of schizophrenia.
* Pregnant or breastfeeding
* Patients with unstable medical conditions
* Patients with previous history of failure to respond to an adequate trial of clozapine
* Patients with a known allergy to risperidone or a previous history of failure to respond to an adequate trial of risperidone. However, patients with known allergies or failure to respond to any of the other medications (aripiprazole, olanzapine, quetiapine or ziprasidone) will not receive that medication if they are randomized to the oral medication arm, but are not excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2006-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina R. Schooler, PhD, Study Director — Steering and Implementation Center
Locations (8):
- United States (8):
  - University of California, Los Angeles, Los Angeles, California
  - Medical College of Georgia, Department of Psychiatry, Augusta, Georgia
  - University of Iowa College of Medicine, Psychiatry Research, Iowa City, Iowa
  - Harvard Medical School -- Massachusetts General Hospital, Boston, Massachusetts
  - Harvard Medical School -- Dr. John C. Corrigan Community Mental Health Center, Fall River, Massachusetts
  - Creighton University, Omaha, Nebraska
  - University of New Mexico, Albuquerque, New Mexico
  - The Zucker Hillside Hospital, Glen Oaks, New York

REFERENCES:
- [Result] Buckley PF, Schooler NR, Goff DC, Hsiao J, Kopelowicz A, Lauriello J, Manschreck T, Mendelowitz AJ, Miller del D, Severe JB, Wilson DR, Ames D, Bustillo J, Mintz J, Kane JM; PROACTIVE Study. Comparison of SGA oral medications and a long-acting injectable SGA: the PROACTIVE study. Schizophr Bull. 2015 Mar;41(2):449-59. doi: 10.1093/schbul/sbu067. Epub 2014 May 27. PMID 24870446

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 357 individuals consented to participation. However, 52 were either ineligible, withdrew consent, or lost to followup. Therefore, 305 individuals were randomized.
Period: Overall Study
Arm/Group | Injectable | Oral
Started | 153 | 152
Completed | 72 | 72
Not Completed | 81 | 80

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Injectable | Oral | Total
Number analyzed (Participants) | 153 | 152 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.18 (11.8) | 38.23 (12.3) | 38.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 42 | 87
  Male | 108 | 110 | 218
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 81 | 78 | 159
  African American | 45 | 40 | 85
  Hispanic | 27 | 31 | 58
  Other | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 153 | 152 | 305
Clinical Global Impressions (CGI) Severity Scale [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impressions Severity Scale is one item completed by a clinician rater. "Considering your total clinical experience with this patient population, how mentally ill is the patient at this time?" The seven possible ratings are as follows.
  1. = Normal, not at all.
  2. = Borderline mentally ill.
  3. = Mildly ill.
  4. = Moderately ill.
  5. = Markedly ill.
  6. = Severely ill
  7. = Among the most extremely ill patients.
  units on a scale | 4.1 (0.84) | 4.0 (0.77) | 4.04 (0.80)

OUTCOME MEASURES:

1. Primary Outcome: Substantial Clinical Deterioration Measured by Psychotic Symptoms
Description: Brief Psychiatric Rating Scale (BPRS) psychosis cluster. Score range is based on the score range for individual items rather than the factor total because is factors have different numbers of items. Score range is 1 -7 where 1 + no symptomatology and 7 = very severe symptoms.
Time Frame: Measured throughout study up to 30 months
Population: We conducted a mixed model regression analysis with two treatment groups X time psychosis cluster scores at each 3 monthly observation from baseline to 30 months. Missing data were treated as MAR
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Injectable | Oral
Number analyzed (Participants) | 153 | 152
units on a scale | 1.8 [1.7 to 1.9] | 2.0 [1.9 to 2.2]

2. Secondary Outcome: Number of Patients Discontinuing From the Study
Time Frame: Measured throughout study up to 30 months
Measure: Number; unit: participants
Arm/Group | Injectable | Oral
Number analyzed (Participants) | 153 | 152
participants | 81 | 80

3. Secondary Outcome: Number of Days in Hospital
Time Frame: Measured throughout study up to 30 months
Population: These data were not collected.
Arm/Group | Injectable | Oral
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Control of Psychiatric Symptoms
Description: Brief Psychiatric Rating Scale (BPRS) total score
Time Frame: Measured throughout study up to 30 months
Population: These data were not collected. No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Injectable | Oral
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Quality of Life Measures
Description: Scale of Functioning (SOF)
Time Frame: Measured throughout study up to 30 months
Population: No data displayed because Outcome Measure has zero total participants analyzed. Data not collected.
Arm/Group | Injectable | Oral
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Side Effects and Metabolic Measures
Description: The highest severity of each of 24 adverse event (AE) that was assessed.over the 30 month study period. The mean severity on a scale of 1 (none) to 4 very severe symptom was recorded at each biweekly visit. Results for each variable are summarized over time so that each subject has a single mean severity rating for each AE. There is no named scale. Each of the side effects measured is named in ways that are clear to medical readers e.g anorexia. The range is 1 none to 4 very severe. Therefore, a higher scale score is worse.
Time Frame: Measured throughout study up to 30 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Injectable | Oral
Number analyzed (Participants) | 143 | 148
units on a scale
  Bruising easily | 1.43 (0.71) | 1.48 (0.75)
  Rash | 1.53 (0.78) | 1.44 (0.71)
  Urticaria (hives, itching) | 1.60 (0.69) | 1.71 (0.84)
  Blurred vision | 1.76 (0.73) | 1.91 (0.83)
  sedation/drowsiness | 2.34 (0.87) | 2.53 (0.78)
  Restlessness | 2.48 (0.76) | 2.43 (0.82)
  Insomnia | 2.38 (0.89) | 2.36 (0.94)
  Malaise (weakness, fatigue) | 2.22 (0.85) | 2.14 (0.87)
  Stiffness | 2.01 (0.82) | 1.97 (0.85)
  Tremor | 1.77 (0.72) | 1.75 (0.80)
  Dizziness | 1.82 (0.79) | 1.78 (0.82)
  Headache | 1.99 (0.88) | 1.89 (0.90)
  Fever | 1.27 (0.49) | 1.24 (0.46)
  Sore Throat | 1.64 (0.78) | 1.57 (0.69)
  Dry Mouth | 2.36 (0.92) | 2.25 (0.94)
  Hypersalivation | 1.76 (0.80) | 1.84 (0.94)
  Enuresis | 1.63 (0.89) | 1.56 (0.83)
  Constipation | 1.75 (0.86) | 1.64 (0.82)
  Diarrhea | 1.65 (0.86) | 1.68 (0.81)
  Anorexia (loss of appetite) | 1.89 (0.86) | 1.69 (0.84)
  Nausea | 1.78 (0.82) | 1.72 (0.80)
  Vomiting | 1.48 (0.72) | 1.51 (0.76)
  Menstrual Irregularity | 1.62 (0.96) | 1.55 (0.86)
  Breast tenderness/galactorrhea | 1.39 (0.69) | 1.32 (0.61)

ADVERSE EVENTS:
Description: 305 participants were randomized. However, 9 never received study medication. Therefore, SAE results are reported for 296 participants. 5 subjects did not have postbaseline AE ratings, and therefore AE results are reported for 291 participants.
Arm/Group | Injectable | Oral
Serious Adverse Events (participants affected / at risk) | 61/146 | 48/150
Other Adverse Events (participants affected / at risk) | 143/143 | 148/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Injectable (N=146) | Oral (N=150)
first relapse often hospitalization (Psychiatric disorders) | 61 | 48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Injectable (N=143) | Oral (N=148)
anorexia (Psychiatric disorders) | 143 | 148 — Anorexia was higher in injectable arm than in oral arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes